CLINICAL TRIAL: NCT05908136
Title: Restoration of the Primary Molars With Strip Crowns and Two Types of Composites
Brief Title: Clinical and Radiographical Evaluation of Two Types of Composite Materialsstrip Crown in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ibraheem Mohammed Mohamed Elshenawe, director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: crowns in pediatric dentistry
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP A (Active Comparator): • Group A: 12 primary molars received stainless steel crowns (SSCs).
  Interventions: Other: restorative materials
- group b (Active Comparator): • Group B: 12 primary molars received resin composite strip crowns (RCSCs).
  Interventions: Other: restorative materials
- group c (Active Comparator): • Group C: 12 primary molars received zirconium-filled composite strip crowns (ZFSCs).
  Interventions: Other: restorative materials

INTERVENTIONS:
Other: restorative materials — two types of composite with strip crown in primary molars
  Other Names: composite materials; strip crown

SUMMARY:
Alterations in oral health of children interfere with their quality of life. Dental caries is the most common public health problem of children . The disease is the result of a complex interaction between acid producing tooth-adherent bacteria and fermentable carbohydrates. Over time, the acids in the dental plaque demineralize enamel and dentin in the fissures and the smooth surfaces of the tooth. The earliest visual sign of dental caries is white spot lesion. If demineralization continues, the surfaces of the white spot will cavitate, resulting in a cavity. If demineralization environment is reduced or eliminated, white spot lesions may remineralize and not progress. Risk factors include high numbers of cariogenic bacteria, high frequency sugar consumption, inadequate salivary flow, insufficient fluoride exposure, poor oral hygiene, and poverty.

The early diagnosis and management of caries still a challenge of dental care for children . The prefabricated metal crowns are often the first choice for the repair of severely damaged primary teeth and have been one of the most effective and efficient methods of tooth restoration in pediatric dentistry since Humphrey first used them in pediatric patients in 1950 . They are used to restore primary or permanent teeth with extensive or multisurface cavities, cervical decalcification, and/or developmental defects .

The prefabricated metal crowns have many advantages over other crown types and dental restorative materials . Their life span is the same as that of an intact primary tooth, they provide protection to the residual tooth structure that may have been weakened after excessive caries removal, the technique sensitivity or the risk of making errors during their application is low and their cost is low .

Despite many advantages, the metal appearance of these crowns is unpleasant to the parents and children and they prefer tooth-colored restorations to silver-colored fillings regardless of location of restorations . Inflammation of the surrounding gingival tissue is a problem frequently associated with prefabricated metal crowns. The incidence of gingivitis has been reported to be higher around poorly fitting crowns than around the crowns considered to be well adapted .

Considering the increasing demand for esthetic restorations, several treatment options have been proposed for primary teeth to overcome this problem such as strip crowns, pre-veneered stainless steel crowns and zirconia crowns .

Strip crown was introduced by Webber et al., in 1979 . strip crowns are available in different brands but the most commonly used resin composite strip crowns worldwide is 3M ESPE crown (3M ESPE Dental). Composite resin strip crowns (SC) have been utilized for over 2 decades to restore carious primary teeth . In spite of a long time of using, there is a paucity of literature concerning the clinical success of these crowns .

Incorporation of ceramic nanofibers in dental composites can significantly improve their mechanical properties and fracture toughness and thus may extend their service life.

This study aimed to assess clinically and radiographicaly of primary teeth restored with stability of the glassionomer and two composite material crown restoration using the preformed strip crown technique in primary molars.

DETAILED DESCRIPTION:
Alterations in oral health of children interfere with their quality of life. Dental caries is the most common public health problem of children . The disease is the result of a complex interaction between acid producing tooth-adherent bacteria and fermentable carbohydrates. Over time, the acids in the dental plaque demineralize enamel and dentin in the fissures and the smooth surfaces of the tooth. The earliest visual sign of dental caries is white spot lesion. If demineralization continues, the surfaces of the white spot will cavitate, resulting in a cavity. If demineralization environment is reduced or eliminated, white spot lesions may remineralize and not progress. Risk factors include high numbers of cariogenic bacteria, high frequency sugar consumption, inadequate salivary flow, insufficient fluoride exposure, poor oral hygiene, and poverty.

The early diagnosis and management of caries still a challenge of dental care for children . The prefabricated metal crowns are often the first choice for the repair of severely damaged primary teeth and have been one of the most effective and efficient methods of tooth restoration in pediatric dentistry since Humphrey first used them in pediatric patients in 1950 . They are used to restore primary or permanent teeth with extensive or multisurface cavities, cervical decalcification, and/or developmental defects .

The prefabricated metal crowns have many advantages over other crown types and dental restorative materials . Their life span is the same as that of an intact primary tooth, they provide protection to the residual tooth structure that may have been weakened after excessive caries removal, the technique sensitivity or the risk of making errors during their application is low and their cost is low .

Despite many advantages, the metal appearance of these crowns is unpleasant to the parents and children and they prefer tooth-colored restorations to silver-colored fillings regardless of location of restorations . Inflammation of the surrounding gingival tissue is a problem frequently associated with prefabricated metal crowns. The incidence of gingivitis has been reported to be higher around poorly fitting crowns than around the crowns considered to be well adapted .

Considering the increasing demand for esthetic restorations, several treatment options have been proposed for primary teeth to overcome this problem such as strip crowns, pre-veneered stainless steel crowns and zirconia crowns .

Strip crown was introduced by Webber et al., in 1979 . strip crowns are available in different brands but the most commonly used resin composite strip crowns worldwide is 3M ESPE crown (3M ESPE Dental). Composite resin strip crowns (SC) have been utilized for over 2 decades to restore carious primary teeth . In spite of a long time of using, there is a paucity of literature concerning the clinical success of these crowns .

Incorporation of ceramic nanofibers in dental composites can significantly improve their mechanical properties and fracture toughness and thus may extend their service life.

This study aimed to assess clinically and radiographicaly of primary teeth restored with stability of the glassionomer and two composite material crown restoration using the preformed strip crown technique in primary molars.

ELIGIBILITY:
Inclusion Criteria:

Primary molars indicated for crown restoration (pulp treated molars indicated for crown

Co-operative child(Frankel scale +ve and ++ve)

The age ranged from 4 to 7 years regardless of sex or socioeconomic background.

Exclusion Criteria:

Badly decayed non-restorable tooth indicated for extraction.

Patients with parafunctional habits like bruxism.

Systemic diseases with oral manifestation or blood diseases.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
fracture and retention score | 6 months
  EXCELLENT GOOD POOR
gingival index | 6 months
  SCORE 0;1;2;3
radiographic pathology | 6 months
  PRESENT OR NOT

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar Univerisity, Cairo, NASR CITY, Egypt

IPD SHARING:
Plan to Share IPD: Yes
PLAN FOR SHARE with other researchers
Supporting Information: Study Protocol, CSR
Time Frame: 6 MONTHS
Access Criteria: NO ACCESS

REFERENCES:
- [Result] Jeong MA, Kim AH, Shim YS, An SY. Restoration of strip crown with a resin-bonded composite cement in early childhood caries. Case Rep Dent. 2013;2013:581934. doi: 10.1155/2013/581934. Epub 2013 Sep 24. PMID 24490090